CLINICAL TRIAL: NCT06313255
Title: A Retrospective Observational Study on the Effects of Probiotics on HBsAg Clearance
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202301-008-1
Record Dates: First submitted 2024-03-10; First posted 2024-03-15 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-03

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Nucleosides

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PegIFNα2b
  Interventions: Drug: PegIFNα2b
- PegIFNα2b+probiotics
  Interventions: Drug: PegIFNα2b+probiotics
- Nucleoside analog
  Interventions: Drug: Nucleoside analog
- Nucleoside analog+probiotics
  Interventions: Drug: Nucleoside analog+probiotics

INTERVENTIONS:
Drug: PegIFNα2b — The patients receive PegIFNα2b therapy
  Groups: PegIFNα2b
Drug: PegIFNα2b+probiotics — The patients receive both PegIFNα2b and probiotics therapy
  Groups: PegIFNα2b+probiotics
Drug: Nucleoside analog — The patients receive nucleoside analog therapy
  Groups: Nucleoside analog
Drug: Nucleoside analog+probiotics — The patients receive both nucleoside analog and probiotics therapy
  Groups: Nucleoside analog+probiotics

SUMMARY:
The goal of this retrospective observational study is to find out the effects of probiotics on HBV clearance. The main question it aims to answer is:

Are the probiotics have an effect in promoting HBV clearance? The participants will observe the HBV clearance rate in chronic hepatitis B patients receive probiotics in addition to the routine antiviral therapy.

Researchers will compare the HBV clearance rate in chronic hepatitis B patients receive probiotics and antiviral therapy with those receiving solely antiviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* chronic hepatitis B patients

Exclusion Criteria:

* patients with malignancies
* patients with other liver diseases
* pregnancy patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is patients with chronic hepatitis B who are receiving antiviral therapy with or without probiotics.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
HBsAg clearance | 48 months

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China